CLINICAL TRIAL: NCT04178928
Title: Can Levothyroxine Treatment Reduce the Development of Cardio-metabolic Disorder in Subclinical Hypothyroidism?
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nashwa Mohamed Abd elwahab, MD candidate, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Sub clinical hypothyroidism
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Subclinical hypothyroïdism
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): patiWill receive L-T4 treatment at a dose 1 µg/kg/day for 12 weeks. And the dose will be titrated every 4 weeksents with SCH will be subjected to clinical, laboratory and imaging assessment and
  Interventions: Drug: Levothyroxine
- Group B (No Intervention): .pWill not receive treatment.atients with SCH will be subjected to clinical, laboratory and imaging assessment and

INTERVENTIONS:
Drug: Levothyroxine — investigate the effect of replacement therapy with levothyroxine on cardiovascular risk factors in children with SCH.
  Arms: group A

SUMMARY:
2. Aim/ Objectives The aim of this study is to evaluate the clinical, laboratory and echocardiographic findings in children with SCH.

To investigate the effect of replacement therapy with levothyroxine on cardiovascular risk factors in children with SCH.

DETAILED DESCRIPTION:
Sub-clinical hypothyroidism (SCH) is a form of thyroid dysfunction in which the thyroid-stimulating hormone (TSH) level is high, while serum total/free thyroxine (T4/fT4) is within the normal reference range . SCH is mostly detected accidentally as most of the patients manifest few or no signs of thyroid dysfunction.

The most common causative factor for SCH is chronic autoimmune thyroiditis characterized by high titers of thyroid peroxidase antibodies, thyroglobulin antibodies and rarely TSH receptor blocking antibodies. However, mutations in several proteins involving in TSH action including TSH receptor gene and mutations of dual oxidase 2 (DUOX2), phosphodiesterase 8B and thyroid peroxidase have also been demonstrated as causes of TSH elevation .

SCH might be associated with endothelial dysfunction due to early changes in proatherogenic profiles as there is elevation in plasma levels of total cholesterol (TC) and low-density lipoprotein-cholesterol (LDL-C) in SCH patients , also there is increased risk of hypertension in SCH patients than in euthyroid .

Many studies found that homocysteine concentration appears to be increased in hypothyroidism and decreased in hyperthyroidism, and there is relationship between hyperhomocysteinemia and cardiovascular disease, including increased platelet aggregation, increased coagulation or reduced thrombolysis and endothelial dysfunction .

The acute-phase reactant hs-CRP is known to be a sensitive and non-specific marker for inflammation, tissue damage and infection . Serum hs-CRP measurements are used to determine cardiovascular risk. hs-CRP is regarded as a predictive marker for myocardial infarction, stroke, peripheral artery disease and sudden cardiac death .

The treatment of children with SCH is controversial; and there is not enough evidence that treatment can prevent the risk of developing cardiovascular and metabolic disorders in SCH.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged from 5-15 years diagnosed with SH (patients with elevated TSH and normal Ft4 on two different measurements 4-6 weeks apart).

Exclusion Criteria:

* 1. Patients with acute or chronic disorders (anemia, infection, diabetes mellitus, malignancy, liver and renal disorder).

  2. Patients with a history of medication that affect thyroid function tests as glucocorticoids, dopamine or dobutamine, amiodarone, lithium, interferons, alemtuzumab.

  3. Patients with BMI>95 percentile.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
: Normalization of TSH. | 12 week
  Normalization of TSH by receive L-T4 treatment at a dose 1 µg/kg/day for 12 weeks. And the dose will be titrated every 4 weeks then check differences in results between baseline assessment and12 weeks after intervention.